CLINICAL TRIAL: NCT06289582
Title: Longitudinal TSPO PET Imaging With [18F]DPA-714 in PPMI (PPMI DPA-714 PET Imaging)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Jonathan E McConathy, M.D. P.h.D., Director for the Division Molecular Imaging and Therapeutics, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R24-004; 022189 (Other Grant/Funding Number: Fox (Michael J.) Foundation for Parkinson's Research)
Record Dates: First submitted 2024-02-13; First posted 2024-03-04 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prodromal and manifest (PD) participants (Experimental)
  Interventions: Drug: [F-18]DPA714 administration IV
- Healthy participants (Experimental)
  Interventions: Drug: [F-18]DPA714 administration IV

INTERVENTIONS:
Drug: [F-18]DPA714 administration IV — brain PET/MRI imaging after [F-18]DPA-714 administration

SUMMARY:
The overall goal of this protocol is to investigate [18F]DPA-714 binding in prodromal and early manifest Parkinson's Disease (PD) and to determine the baseline and change from baseline in [18F]DPA-714 binding in PD participants during a 24-month interval.

Primary Objectives

* To compare [18F]DPA-714 binding in prodromal and manifest PD and healthy volunteers.
* To determine the longitudinal change in [18F]DPA-714 during a 24-month interval for prodromal and early initially untreated PD participants.

Secondary Objectives

* To evaluate the correlation between baseline [18F]DPA-714 and PPMI clinical and biomarker outcomes.
* To evaluate the correlation between the longitudinal change of [18F]DPA-714 and PPMI clinical and biomarker outcomes
* To acquire safety data following injection of [18F]DPA-714

ELIGIBILITY:
Inclusion Criteria:

* A prodromal PD and Healthy participant enrolled in PPMI Clinical protocol
* A PD participant enrolled in PPMI Clinical protocol who has not started symptomatic treatment at time of enrollment or in the first 2 years of participation.
* Able to provide informed consent
* Must have screening genetic testing documenting high binder at the at the known TSPO gene polymorphism (rs6971)
* Male or Female (Females must meet additional criteria specified below, as applicable)

  • Females must be of non-childbearing potential or using a highly effective method of birth control 14 days prior to until at least 24 hours after injection of [18F]DPA-714
* Non-childbearing potential is defined as a female that must be either postmenopausal (no menses for at least 12 months prior to PET scan) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy).
* Highly effective method of birth control is defined as practicing at least one of the following: A birth control method that results in a less than 1% per year failure rate when used consistently and correctly, such as oral contraceptives for at least 3 months prior to injection, an intrauterine device (IUD) for at least 2 months prior to injection, or barrier methods, e.g., diaphragm or combination condom and spermicide. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) is not acceptable.

  * Females of childbearing potential must not be pregnant, breastfeeding or lactating.
  * Includes a negative urine pregnancy test prior to injection of [18F]DPA-714 on day of PET scan.

Exclusion Criteria:

* Exposure to a total effective dose equivalent of 50 millisievert (mSv) for the whole body, which is the annual limit established by the US Code of Federal Regulations , during the past year.
* Any other medical or psychiatric condition or lab abnormality, which in the opinion of the Site Investigator might preclude participation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Measure baseline and follow up regional brain TSPO levels using [18F]DPA-714-PET in prodromal PD. | 24 months
  The changes over time in neuroinflammation based on TSPO will be assessed by comparing TSPO-PET imaging at baseline, 12 months and 24 months after enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan McConathy, MD, PhD, Principal Investigator — University of Alabama at Birmingham; David Standaert, MD, PhD, Study Director — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No